CLINICAL TRIAL: NCT02209168
Title: Differences in Ovarian Reserve Markers, Vitamin D Serum Levels and Reproductive Outcomes Between Infertile Indian, Arabian and Caucasian Population
Brief Title: Differences in Ovarian Reserve Markers and Vitamin D Between Infertile Indian, Arabian and Caucasian Population
Status: Withdrawn | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, Carlos Iglesias, MD, IVI Madrid
Other Study IDs: 1405-MAD-020-JG
Record Dates: First submitted 2014-06-27; First posted 2014-08-05 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve; Vitamin D Deficiency; Hormone Deficiency; Follicular Cyst of Ovary
Keywords: AMH, ACF, VIT D, Ethnicity
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vitamine D serum levels.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Infertile Indian Population: 200 Infertile Indian population
- Infertile arabian population: 200 Infertile Arabian population
- Infertile caucasian population: 200 Infertile Caucasian population

SUMMARY:
The aim of this study is to confirm the difference in ovarian reserve markers and serum vitamine D levels between infertile indian, arabian and caucasian population.

DETAILED DESCRIPTION:
200 caucasian, indian, and arab patients

ELIGIBILITY:
Inclusion Criteria:

WOMEN BETWEEN 21-43 YEARS FIRST OR SECOND IN VITRO FERILIZATION TREATMENT DUE TO TUBAL, MASCULINE OR PREVIOUS INTRAUTERINE INSEMINATION FAIL TREATMENT

Exclusion Criteria:

POLYCYSTIC PATIENTS ENDOMETRIOSIS GRADE III OR IV INFLAMMATORY PELVIC DISEASE

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: WOMEN BETWEEN 21-43 YEARS FIRST OR SECOND IN VITRO FERTILIZATION TREATMENT DUE TO TUBAL, MASCULINE OR PREVIOUS INTRAUTERINE INSEMINATION FAIL TREATMENT
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve markers: antimullerian hormone, FSH, antral follicle count | beginning of the treatment cycle

SECONDARY OUTCOMES:
Serum vitamin D levels | Beginning of their treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS IGLESIAS, MD, Principal Investigator — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Spain